CLINICAL TRIAL: NCT02803710
Title: Prevalence of Enterobacteriaceae With Decreased Susceptibility to Carbapenems in Eastern Inter- Region
Brief Title: Prevalence of Enterobacteria With Decreased Susceptibility to Carbapenems in Eastern Inter- Region
Acronym: CARBAFREST
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CHU de Reims (Other)
Responsible Party: Sponsor
Other Study IDs: PR11006
Record Dates: First submitted 2016-06-08; First posted 2016-06-17 (Estimated); Last update posted 2016-06-20 (Estimated); Status verified 2016-06

CONDITIONS: Infection With Beta-lactam Resistance in Enterobacteriaceae

STUDY DESIGN:
Observational Model: Case-Control

GROUPS / COHORTS (2):
- Case group: patients with decreased susceptibility to carbapenems Enterobacteriaceae isolate
  Interventions: Other: Microbiological study
- Control-group: patients with Enterobacteriaceae isolate without decreased susceptibility to carbapenems
  Interventions: Other: Microbiological study

INTERVENTIONS:
Other: Microbiological study

SUMMARY:
Upon penicillins' introduction, inactivation of beta- lactam antibiotics by enzymes produced by bacteria was demonstrated. Until recently, carbapenems were a relatively spared subclass by these enzymes which makes the molecules of last resort in serious infection. Recently the prevalence of enzymes hydrolysing carbapenem, the carbapenemases, was increasing in some countries. But these carbapenemases are not the only mechanism involved in a decreased susceptibility to carbapenems which is sometimes linked to the conjunction of several resistance mechanisms. Data available on the epidemic situation of this new resistance are essential for improving their detection, the management of infections in patients and prevent the occurrence of epidemic. In this context, the investigators propose a study in the North-East inter-region to estimate the prevalence of Enterobacteriaceae with decrease susceptibility to carbapenems and look for risk factors for infection with this type of bacteria. The study is conducted in five teaching hospitals (Besançon, Dijon, Nancy, Reims and Strasbourg) and two general hospitals (Colmar and Troyes) in North-Eastern France. For one year, all the Enterobacteriaceae isolates with a decreased susceptibility to carbapenems (CDSE) according to the 2012 Antibiogram Comity of the French Microbiology Society (CA-SFM) (MIC of ertapenem > 0.5 μg/mL) are collected and sent to the bacteriology laboratory of the Reims University Hospital. Among these strains 105 are randomly selected. The clinical study is conducted as follow: for each patient with CDSE isolate included in a center, 2 control patients are selected. They are the patients having the 2 Enterobacteriaceae isolates, with no reduced susceptibility to carbapenems and following the CDSE isolate in the same center.

Microbiological study : identification of isolates is performed using MALDI-TOF (Bruker Daltonics, Bremen, Germany). Antibiotic susceptibilities is determined by the disc diffusion method according to European Committee on Antimicrobial Susceptibility Testing (EUCAST) guidelines (www.EUCAST.org) and extended-spectrum beta-lactamase (ESBLs) are detected by the double-disc synergy test and carbapenem minimal inhibitory concentrations (MICs to Imipenem, Ertapenem, Doripenem and Meropenem) determined using E-test® strips. Metallo-β-lactamase production was screened with the MβL Etest (bioMérieux, Marcy l'Etoile, France). Beta-lactamases detected using polymerase chain reaction (PCR). Carbapenemase-encoding genes (blaKPC, blaVIM, blaIMP, blaNDM, blaOXA-23-like, blaOXA-24-like, blaOXA-58-like and blaOXA-48-like) were screened using multiplex PCRs and blaIMI and blaGES with simplex PCRs. All the blaOXA-48-like detected were subsequently sequenced. Genes blaTEM, blaSHV, blaCTX-M and blaOXA were detected by PCR using specific primers. Plasmid-mediated AmpC-type genes blaACC, blaFOX, blaMOX, blaDHA, blaCMY and blaMIR were screened using multiplex PCRs. All the beta-lactamases are sequenced. Mutations in the quinolone resistance determining region (QRDR) are identified by PCR and sequencing in the gyrA, gyrB, parC and parE genes. Qnr and qepA genes are detected by real-time PCR, aac(6')-Ib-cr by pyrosequencing and oqxAB by conventional PCR. Genotyping is performed with pulsed-field gel electrophoresis (PFGE) and multilocus sequence typing (MLST).

Statistical analysis : qualitative variables are analysed with the Chi2 test and the two-tailed Fisher exact test. Quantitative variables are compared using the Mann-Whitney test. Then, a multivariate analysis is conducted: logistic regression with stepwise factors as explanatory variables with p <0.20 in the univariate analysis as input threshold and output set at 0.20.The results are considered statistically significant when P < 0.05.

Expected results : this study will give the proportion of the different species involved, of the carbapenemase in comparison to the other mechanisms, the level of resistance in MIC. Risk factors such as previous antibiotic treatment, underlying disease severity or clonal strain transmission will be evidenced, allowing to identify prevention control measure to implement.

ELIGIBILITY:
Inclusion Criteria:

* Cases: patients (infected or colonized) with an Enterobacteriaceae isolate with decreased susceptibility to carbapenems
* Controls: patients (infected or colonized) with an Enterobacteriaceae isolate not having reduced susceptibility to carbapenems and for which the strain was isolated following an Enterobacteriaceae isolate with decreased susceptibility to carbapenems (2 controls per case).

Exclusion Criteria:

* <18yo

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For one year, all the Enterobacteriaceae isolates with a decreased susceptibility to carbapenems (CDSE) according to the 2012 Antibiogram Comity of the French Microbiology Society (CA-SFM) (MIC of ertapenem > 0.5 μg/mL) are collected and sent to the bacteriology laboratory of the Reims University Hospital. Among these strains 105 are randomly selected. The clinical study is conducted as follow: for each patient with CDSE isolate included in a center, 2 control patients are selected. They are the patients having the 2 Enterobacteriaceae isolates, with no reduced susceptibility to carbapenems and following the CDSE isolate in the same center.
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Antibiotic susceptibilities by the disc diffusion method | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Reims, Reims, France

REFERENCES:
- [Result] Guillard T, Cholley P, Limelette A, Hocquet D, Matton L, Guyeux C, Lebreil AL, Bajolet O, Brasme L, Madoux J, Vernet-Garnier V, Barbe C, Bertrand X, de Champs On Behalf Of CarbaFrEst Group C. Fluoroquinolone Resistance Mechanisms and population structure of Enterobacter cloacae non-susceptible to Ertapenem in North-Eastern France. Front Microbiol. 2015 Oct 23;6:1186. doi: 10.3389/fmicb.2015.01186. eCollection 2015. PMID 26557115
- [Result] Liapis E, Pantel A, Robert J, Nicolas-Chanoine MH, Cavalie L, van der Mee-Marquet N, de Champs C, Aissa N, Eloy C, Blanc V, Guyeux C, Hocquet D, Lavigne JP, Bertrand X; ONERBA. Molecular epidemiology of OXA-48-producing Klebsiella pneumoniae in France. Clin Microbiol Infect. 2014 Dec;20(12):O1121-3. doi: 10.1111/1469-0691.12727. Epub 2014 Jul 29. PMID 24942039